CLINICAL TRIAL: NCT01484041
Title: A Phase I/II Trial of TKI258 (Dovitinib) in Combination With an Aromatase Inhibitor in Patients With Metastatic Breast Cancer
Brief Title: Dovitinib Plus an Aromatase Inhibitor for Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Decision by company to cease development of dovitinib
Sponsor: Georgetown University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 2010-535
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2015-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; postmenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one; Aromatase Inhibitors; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dovitinib plus aromatase inhibitors (Experimental): Dovitinib with aromatase inhibitor
  Interventions: Drug: Dovitinib; Drug: Aromatase Inhibitors

INTERVENTIONS:
Drug: Dovitinib — Dovitinib at the recommended Phase 2 dose for 5 consecutive days followed by a 2-day rest
  Other Names: TKI258
Drug: Aromatase Inhibitors — Patients will receive one of the aromatase inhibitors either anastrozole 1 mg po daily, letrozole 2.5 mg po daily, or exemestane 25 mg po daily
  Other Names: Arimidex; Femara; Aromasin

SUMMARY:
This study is for women with confirmed hormone receptor positive HER-2 negative advanced breast cancer with evidence of disease resistance to an aromatase inhibitor.

The purpose of this study is to determine how well these medications work together and/or if they have any side effects in patients with hormone-receptor positive metastatic breast cancer who have demonstrated progression of disease after first line hormonal therapy.

This research is being done to determine if taking an already approved medicine (aromatase inhibitor) in combination with a new medication (dovitinib) results in better outcomes for patients with this disease.

Both dovitinib and an aromatase inhibitor are pills that will be taken at home.

DETAILED DESCRIPTION:
This is a Phase I/Phase II open-label single arm trial of dovitinib in combination with anastrozole 1 mg daily, exemestane 25 mg daily, or letrozole 2.5 mg daily. Study subjects will receive the aromatase inhibitor on which they had previously derived clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with breast cancer either in the primary or metastatic setting
* Tumor must be estrogen receptor and/or progesterone receptor positive and Her-2 negative
* Evidence of disease resistance to an aromatase inhibitor
* ECOG performance status 0 or 1
* Age 18 years or older
* Adequate laboratory values
* Able to give written informed consent
* Measurable disease
* No more than 2 prior chemotherapy regimens in the metastatic setting
* Unlimited prior hormonal therapy in the metastatic setting
* Life expectancy of greater than 3 months
* Post-menopausal
* Tumor must be available for central testing for FGFR1 amplification by FISH/CISH

Exclusion Criteria:

* Brain metastases
* Another primary malignancy within 3 years prior to starting drug therapy with the exception of adequately treated in-site carcinoma of the uterine cervix or skin cancer
* Chemotherapy within 3 weeks prior to starting study drug or not recovered from side effects of previous therapy
* Administration of nitrosurea or mitomycin-C within 6 weeks prior to starting study drug or not recovered from side effects of such therapy
* Administration of biologic therapy within 6 weeks prior to starting study drug or not recovered from side effects of such therapy
* Radiotherapy within 4 weeks prior to starting study drug or 2 weeks in the case of localized radiotherapy or not recovered from radiotherapy toxicities
* major surgery, open biopsy or significant traumatic injury within 4 weeks prior to starting study drug or a minor procedure, percutaneous biopsy or placement of a vascular access device within 1 week prior to starting study drug or not recovered from side effects of such procedure or injury
* Chronic concomitant bisphosphonate therapy for the prevention of bone metastases. Bisphosphonate/ denosumab therapy for the management of bone metastases or for the treatment of osteoporosis s allowed.
* Impaired cardiac function or clinically significant cardiac disease
* Impairment of GI function or GI disease that may significantly alter the absorption of dovitinib
* Cirrhosis, chronic active hepatitis, or chronic persistent hepatitis
* Known diagnosis of HIV infection
* Anticoagulation treatment with therapeutic doses of warfarin
* Any concurrent severe and/or uncontrolled concomitant medical condition that could cause unacceptable safety risks or compromise compliance with the protocol
* Pregnant or breast-feeding
* Unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Isaacs, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Will not be reporting outcome data as study closed by sponsor prior to completing accrual. Will be reporting aggregate findings for correlative science project

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dovitinib Plus Aromatase Inhibitors
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dovitinib Plus Aromatase Inhibitors
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 53.5 [32 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate
Description: Complete response, partial response, or stable disease at 24 weeks from trial entry as per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Dovitinib Plus Aromatase Inhibitors
Number analyzed (Participants) | 12
participants | 1

2. Secondary Outcome: Recommended Phase 2 Dose
Description: The dose of dovitinib at which 1 or less subjects experience a dose limiting toxicity when administered every day for 5 days followed by 2 days off schedule in combination with an aromatase inhibitor
Time Frame: 4 weeks
Population: Subjects on study evaluated for toxicity
Measure: Number; unit: mg
Arm/Group | Dovitinib Plus Aromatase Inhibitors
Number analyzed (Participants) | 6
mg | 400

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants experiencing adverse events
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Dovitinib Plus Aromatase Inhibitors
Number analyzed (Participants) | 12
participants | 12

4. Secondary Outcome: Pharmacodynamic Effects
Description: Expression of pFGFR, pFRS2, pERK in tumor tissue and VEGF, bFGF, PLGF, sVEGFR1/2 and FGF23 levels in plasma
Time Frame: 24 weeks
Population: Data were not collected for this outcome
Arm/Group | Dovitinib Plus Aromatase Inhibitors
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-free Survival
Description: Length of time from study entry until progressive disease
Time Frame: 24 weeks
Population: Data not collected for this outcome as study terminated by company prior to completing accrual
Arm/Group | Dovitinib Plus Aromatase Inhibitors
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Dovitinib Plus Aromatase Inhibitors
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dovitinib Plus Aromatase Inhibitors (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dovitinib Plus Aromatase Inhibitors (N=12)
Diarrhea (Gastrointestinal disorders) | 8 (14)
Nausea (Gastrointestinal disorders) | 9 (11)
Vomiting (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 6 (11)
Hot flashes (Endocrine disorders) | 4 (14)
Pain (Musculoskeletal and connective tissue disorders) | 6 (14)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Thromboembolism (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (2)
Headache (Nervous system disorders) | 3 (3)
Dehydration (General disorders) | 3 (4)
Dizziness (Nervous system disorders) | 1 (1)
Edema (Blood and lymphatic system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (3)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (2)
Alanine aminotransferase increased (Hepatobiliary disorders) | 6 (10)
Creatinine increased (Renal and urinary disorders) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4)
Platelet decreased (Blood and lymphatic system disorders) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (8)
White blood cell count decreased (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No